CLINICAL TRIAL: NCT05105568
Title: Process-Based Therapy in an Outpatient Setting: A Multiple Baseline Study
Brief Title: Process-Based Therapy in an Outpatient Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moved to different institution and continuing was not feasible.
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6214
Record Dates: First submitted 2021-10-05; First posted 2021-11-03 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Nonconcurrent multiple baseline design with three dyads.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Process-based therapy (Experimental)
  Interventions: Behavioral: Process-based therapy

INTERVENTIONS:
Behavioral: Process-based therapy — Process-based therapy (PBT) is a meta-theoretical model of evidence-based therapies that organizes adaptive and maladaptive processes of change using complex and dynamic networks based on an evolution science framework. Depending on the participant's presentation, PBT would be shaped by different evidence-based techniques. Examples of evidence-based procedures include: behavioral activation, exposures, mindfulness, self-compassion, values exploration, and contingency management.

SUMMARY:
The proposed study aims to examine the effects of process-based therapy on 6 adult patients presenting for treatment at a university community outpatient clinic using a nonconcurrent multiple baseline design.

DETAILED DESCRIPTION:
Process-based therapy (PBT) is a meta-theoretical model of evidence-based therapies that organizes adaptive and maladaptive processes of change using complex and dynamic networks based on an evolution science framework. Although papers and books have been written on PBT, PBT has yet to be empirically tested as an intervention in a clinical setting. The proposed study aims to examine the effects of PBT on 6 adult patients presenting for treatment at a university community outpatient clinic using a nonconcurrent multiple baseline design. We hypothesize that network structures of patients will change in an adaptive direction over the course of PBT and that these changes will be maintained at 1-month follow-up.

The study will take place remotely over HIPAA-compliant Zoom or in person at the Center for Anxiety and Related Disorders (CARD), depending on the status of the COVID-19 pandemic and participants' preferences. Variables of interest include idiographic items specific to the individual (e.g., treatment goals, problem behaviors, valued action, psychological phenomena, contextual influences) and physiological data (e.g., physical activity, screen time). Throughout the study until 1-month follow-up, participants will be randomly prompted 4 times a day to rate idiographic items via Ethica, an app-based platform for smartphones that collects questionnaire data and passive objective data from sensors. Physiological data will be collected passively through Ethica. These variables will comprise the network used to characterize each participant's presentation. In addition to examining network structures, we will use the Process-Based Assessment Tool (PBAT; Ciarrochi, Hayes, Hofmann, 2021) as a nomothetic measure of PBT-related improvement. The proposed study will provide a proof of concept for PBT, evaluate its efficacy, and demonstrate how it can be applied in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to provide written informed consent
2. Ability to sufficiently communicate in English as assessed through phone screening and the ability to answer study questionnaires
3. At least 18 years old
4. Seeking psychological treatment at CARD (participants do not need to meet criteria for a specific Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition diagnosis)
5. Willingness to abstain from other psychotherapies for duration of study (up to 1-month follow-up; this is so we can be more confident that changes observed during the study are attributable to the study intervention rather than an external intervention; clinically, it is also typically counterproductive for a patient to see multiple therapists at the same time)
6. Working smartphone with internet connection
7. Stable on current psychotropic medications (or off medication for 2 weeks)
8. If participating remotely, access to private room where they will not be disturbed during study sessions

Exclusion Criteria:

1. Suicidality (ideation, intent, or specific plan) significant enough to require higher level of care than outpatient, as determined by CARD phone screening (patients on the CARD waitlist who comprise our recruitment pool are prescreened), the Mini International Neuropsychiatric Interview (MINI), or otherwise determined by the Investigator
2. Currently receiving another psychological treatment
3. Active psychosis, mania, or significant personality dysfunction as assessed through CARD phone screening (patients on the CARD waitlist who comprise our recruitment pool are prescreened), the MINI, or otherwise determined by the Investigator
4. Serious neurological impairment as assessed through phone screening items or otherwise determined by the Investigator
5. Any other reason as determined by the Investigator which may lead to an unfavorable risk-benefit of study participation, interfere with study compliance, or confound study results

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Individual network structure | Up to 7 months
  Network models will be created using intensive longitudinal data collected four times daily. Variables to be measured will depend on the participant's presenting concern. For example, if Participant A reports struggling with avoiding work meetings related to fears about how they will be perceived by their supervisor and co-workers, then we might track percentage of work meetings attended (behavioral goal) and fear of social evaluation (source of distress). Where possible, these items will be assessed using a visual analog scale ranging from 0 to 100 to ensure an adequate range of responding. Because items will be personalized to the participant's presenting concern, we will not be using a standardized scale or questionnaire. Rather, we will be developing idiographic items specific to the participant's presentation and assess variables relevant to the individual.

SECONDARY OUTCOMES:
Process-Based Assessment Tool | Up to 7 months
  The Process-Based Assessment Tool (PBAT) is a new measure that is currently being validated (Ciarrochi et al., 2021, in preparation). The PBAT has 9 subscales: affect, cognitive processes, attention, social/connection needs, motivation/autonomy needs, overt behavior/competence needs, health, variation, and retention.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Anxiety and Related Disorders (CARD), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciarrochi, J., Hayes, S. C., & Hofmann, S. G. (2021). Assessing processes of change in psychological interventions: The Process-Based Assessment Tool (PBAT). Manuscript in preparation. Institute for Positive Psychology and Education, Australian Catholic University.
- [Background] Hofmann, S. G., Hayes, S. C., & Lorscheid, D. N. (2021). Learning process-based therapy: A skills training manual for targeting the core processes of psychological change in clinical practice. New Harbinger.